CLINICAL TRIAL: NCT02782065
Title: Validation Of The Hospital Asthma Severity Score (HASS) In Children Ages 2-18 Years Old
Brief Title: Validation of the Hospital Asthma Severity Score (HASS)
Acronym: HASS
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Leah Abecassis, Nurse Practice Specialist, Boston Children's Hospital
Other Study IDs: P00022204
Record Dates: First submitted 2016-05-06; First posted 2016-05-25 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Asthma
Keywords: validation; pediatrics; asthma severity
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric patients with Asthma: 165 patients aged 7 to 18 years, and 30 patients aged 2 to 6 years
  Interventions: Other: Not an interventional study

INTERVENTIONS:
Other: Not an interventional study

SUMMARY:
The purpose of this research will be to evaluate the reliability and validity of the HASS tool in a cohort of patients' ages 7 to18 years old against the gold standard of spirometry, and in ages 2 to 6 against spirometry, if possible, and the most similar validated tool, the PRAM.

DETAILED DESCRIPTION:
Children aged 7-18 years will have a HASS score obtained by two providers. After scoring is complete, a pulmonary technician will perform the spirometry test.

Children aged 2 to 6 years old will concurrently (but separately) have their asthma severity graded by 2 individual measurers using the HASS tool and the PRAM tool. If consented to perform spirometry, this test will be performed after the tool(s) scores have been obtained.

The spirometry tests will be interpreted by a board-certified pediatric pulmonologist.

Descriptive statistics will be used for preliminary analysis to describe the sample characteristics, outliers, and representativeness of the data.

Primary Aim 1. To describe the inter-rater reliability for the HASS as scored by 2 individual health care providers Data Analysis 1. Use of an overall percentage of agreement, weighted and unweighted kappa and the intraclass correlation coefficient will show the inter-rater reliability of the HASS tool. For each measure, percent agreement between raters and Cohen's kappa statistic (rater agreement adjusted for chance agreement) will be reported.

Primary Aim 2. To evaluate construct validity of the HASS tool in a cohort of patients' ages 7 to18 years old as compared to forced expiratory volume through spirometry

Data Analysis 2. Treating the outcomes as continuous, a correlation coefficient will be computed for HASS and %Forced Expiratory Volume 1. Sub-analyses will also be performed by age group and by %Forced Expiratory Volume1 severity level to see whether the correlation of HASS and %Forced Expiratory Volume1 is consistent across age and asthma severity strata. Treating the outcomes as categorical, if the HASS and %Forced Expiratory Volume1 are each categorized into three levels (mild, moderate, severe), then the investigator could classify each of the nine cells of a 3 by 3 table (HASS X %Forced Expiratory Volume1) as either:

1. concordant (three cells; complete agreement: both tests say 'Severe', for instance),
2. discordant (four cells; e.g. one test says Moderate while the other say Mild) and
3. grossly discordant (two cells; one test says Severe when the other says Mild). For the Receiver Operating Curve analysis, the Forced Expiratory Volume will be dichotomized as Severe (%Forced Expiratory Volume1<60% predicted) versus Less Severe (%Forced Expiratory Volume1≥60% predicted). In analyzing these data, the correlation (continuous), 3 by 3 table (categorical), and Receiver Operating Curve (dichotomous %Forced Expiratory Volume1) treatments will be presented, with the continuous result considered primary. A high level of agreement is expected between the HASS and the spirometry severity score to make the case that the HASS can be used in place of the %Forced Expiratory Volume1 test.

Secondary Aim 3. To evaluate construct validity of the HASS tool in a cohort of patients' ages 2 to 6 years old as compared to forced expiratory volume through spirometry.

Data Analysis 3. Treating the outcomes as continuous, a correlation coefficient will be computed for HASS and %Forced Expiratory Volume1. Treating the outcomes as categorical, if the HASS and %Forced Expiratory Volume1 are each categorized into three levels (mild, moderate, severe), then the investigator could classify each of the nine cells of a 3 by 3 table (HASS X %Forced Expiratory Volume1) as concordant, discordant or grossly discordant (as described in Data Analysis 2). An adequate level of observed agreement would be 80% of observations in agreement cells, 18% discordant, and 2% in grossly discordant cells. In analyzing these data, both the correlation (continuous) and 3 by 3 table (categorical) treatments will be presented, with the continuous result considered primary. A high level of agreement is expected between the HASS and the spirometry severity score to make the case that the HASS can be used in place of the spirometry.

Secondary Aim 4. To evaluate construct validity of the HASS tool in a cohort of patients' ages 2 to 6 years old as compared to the Preschool Respiratory Assessment Measure (PRAM) Data Analysis 4. Treating the outcomes as continuous, a correlation coefficient will be computed for HASS and PRAM. If the HASS and PRAM are each categorized into three levels (mild, moderate, severe), then the investigator could classify each of the nine cells of a 3 by 3 table (HASS X PRAM) as either concordant, discordant, or grossly discordant (as described in Data Analysis 2). An adequate level of observed agreement would be 80% of observations in agreement cells, 18% discordant, and 2% in grossly discordant cells.

ELIGIBILITY:
Inclusion Criteria:

* asthma exacerbation

Exclusion Criteria:

* continuous albuterol and/or
* pneumonia, croup, varicella, cystic fibrosis, broncho-pulmonary dysplasia, cardiac or kidney disease AND
* previously approached for participation in the study

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with asthma exacerbation in the emergency room, inpatient medical units, and medicine intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leah Abecassis, MSN, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Childrens Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
To ensure anonymity and confidentiality of participants, the investigators will not be sharing individual data. A summary report will be provided to participants upon request.

REFERENCES:
- [Derived] Abecassis L, Gaffin JM, Forbes PW, Schenkel SR, McBride S, DeGrazia M. Validation of the Hospital Asthma Severity Score (HASS) in children ages 2-18 years old. J Asthma. 2022 Feb;59(2):315-324. doi: 10.1080/02770903.2020.1852414. Epub 2020 Dec 2. PMID 33198536

RESULTS

PARTICIPANT FLOW:
Groups:
- Pediatric Patients With Asthma: 34 patients aged 7 to 18 years, and 24 patients aged 2 to 6 years
  Not an interventional study
Period: Overall Study
Arm/Group | Pediatric Patients With Asthma
Started | 58
Completed | 58
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pediatric Patients With Asthma
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 58
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 9
Race/Ethnicity, Customized [Number; unit: participants] — Population: There were two participants classified as two different races, and one participant had missing data for that question. With those extra 2 added and 1 not included, it would bring the total number in the race table to be 59.
  participants
    Caucasian: number analyzed (Participants) | 57
    Caucasian | 17
    Black/African American: number analyzed (Participants) | 57
    Black/African American | 24
    Asian: number analyzed (Participants) | 57
    Asian | 2
    Dominican: number analyzed (Participants) | 57
    Dominican | 3
    Other: number analyzed (Participants) | 57
    Other | 4
    Unknown: number analyzed (Participants) | 57
    Unknown | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Inter-rater Reliability for the Hospital Asthma Severity Score (HASS)
Description: The inter-rater reliability (the percent of agreement among raters) for the HASS as scored by 2 individual health care providers. Inter-rater agreement refers to the agreement between the single clinician who was Rater 1 and the second clinician rating the patient (Rater 2), regardless of which clinician served as Rater 2
Time Frame: 4 years and 9 months
Measure: Number; unit: percentage of agreement between raters
Arm/Group | Pediatric Patients With Asthma
Number analyzed (Participants) | 58
percentage of agreement between raters | 29

2. Primary Outcome: Inter-rater Reliability for the Pediatric Respiratory Assessment Measure (PRAM)
Description: The inter-rater reliability for the PRAM as scored by 2 individual health care providers. Inter-rater agreement refers to the agreement between the single clinician who was Rater 1 and the second clinician rating the patient (Rater 2), regardless of which clinician served as Rater 2.
Time Frame: 4 years and 9 months
Measure: Number; unit: percentage of agreement between raters
Arm/Group | Pediatric Patients With Asthma
Number analyzed (Participants) | 58
percentage of agreement between raters | 28

3. Primary Outcome: Intra-rater Reliability Between HASS and PRAM
Description: The intra-rater reliability between HASS and PRAM as scored by 2 individual health care providers. Intra-rater agreement refers to the with-in rater agreement between the PRAM and HASS categorical ratings. This was calculated separately for Rater 1 and Rater 2. The intra-rater agreement for Rater 2 was calculated by pooling the data from the Rater 2 clinicians.
Time Frame: 4 years and 9 months
Measure: Number; unit: percentage of agreement between raters
Arm/Group | Pediatric Patients With Asthma
Number analyzed (Participants) | 58
percentage of agreement between raters
  Rater 1 | 71
  Rater 2 | 64

4. Primary Outcome: Correlation Between the HASS and Forced Expiratory Volume in 1 Second (FEV1)
Description: The correlation coefficient between the HASS tool and FEV1 measurements.
Time Frame: 4 years, 9 months
Population: There were 29 patients out of 58 that performed spirometry and therefore were able to be analyzed for this data.
Measure: Number; unit: correlation coefficient
Groups:
- Pediatric Patients With Asthma: 29 patients aged 2 to 18 years
  Not an interventional study
Arm/Group | Pediatric Patients With Asthma
Number analyzed (Participants) | 29
correlation coefficient | -.31

5. Primary Outcome: Correlation Between the PRAM and FEV1
Description: The correlation between the PRAM and FEV1
Time Frame: 4 years 9 months
Population: There were 29 patients out of 58 that performed spirometry and therefore were able to be analyzed for this data.
Measure: Number; unit: correlation coefficient
Arm/Group | Pediatric Patients With Asthma
Number analyzed (Participants) | 29
correlation coefficient | -.30

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at a single point in time during the data collection (approximately 30 minutes).
Arm/Group | Pediatric Patients With Asthma
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT02782065/Prot_SAP_000.pdf